CLINICAL TRIAL: NCT06519474
Title: Effect of Elastic Chest Compression on Functional Exercise Capacity and Respiratory Performance in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202405096RINE
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: COPD; Hyperinflation
Keywords: chronic obstructive pulmonary disease; dynamic hyperinflation; elastic chest compression; functional exercise capacity; respiratory performance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper chest compression (Experimental): The Theraband will be wrapped around the subject's upper chest with upper edge of the Theraband aligned to the 3rd intercostal space and fastened on the upper rib cage for the upper chest compression arm.
  Interventions: Device: Theraband chest compression
- Lower chest compression (Experimental): The Theraband will be wrapped around the subject's lower rib cage by placing the central horizontal part of the Theraband at the xiphoid process of the sternum for the lower chest compression arm.
  Interventions: Device: Theraband chest compression

INTERVENTIONS:
Device: Theraband chest compression — Chest compression applicated via a Red Theraband over the upper or lower chest region

SUMMARY:
The goal of this clinical trial is to investigate the effects of elastic chest compression on functional exercise capacity and respiratory performance of patients with COPD. The main questions it aims to answer are:

Is there difference in functional exercise capacity and respiratory performance without or with the use of elastic upper chest compression? Is there difference in functional exercise capacity and respiratory performance between the use of elastic upper chest compression and elastic lower chest compression?

Participants will:

Be evaluated under three conditions on three different days: without elastic compression, with upper chest compression, and with lower chest compression, with the order of compression application randomly assigned.

The functional capacity and respiratory muscle performance of all patients will be evaluated.

The days for evaluation will be at least three days apart from each other.

DETAILED DESCRIPTION:
Participants will be evaluated under three conditions: without elastic compression, with upper chest compression, and with lower chest compression, with the order of compression application randomly assigned. A Red Theraband will be used to apply compression to the upper and lower regions of the chest. For a standardized approach to apply compression, the top edge will be aligned with the 3rd intercostal space for the upper chest compression, while the central horizontal part will line up with the xiphoid process of the sternum for the lower chest compression. After exhaling to the EELV, the circumferences of the upper and lower chest regions will be measured, using the 3rd intercostal space as the measurement mark for the upper chest and the xiphoid process of the sternum as the measurement marks for the lower chest. The Thera-Band will be adjusted to 90% of the measured circumferences, ensuring it is securely fastened and standardized resistance is applied consistently to the thoracic regions of interest throughout the study. After chest compression is applied, participants will undergo measurements for functional exercise capacity and respiratory muscle performance.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years old
* has a clinical diagnosis of COPD without infection or acute exacerbation in the previous four weeks
* is capable of cooperating with the required tests and measurements of the study

Exclusion Criteria:

* has any clinical diagnosis that could affect test outcomes (e.g., neuromyopathy)
* has experienced unstable angina or an acute myocardial infarction within the last month
* has adjusted COPD related medication within the last month
* a Mini-Mental State Examination (MMSE) score below 24

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | up to 3 weeks
  6 minute walk test measured in meters
Respiratory muscle performance | up to 3 weeks
  Maximum inspiratory (MIP) and expiratory pressures (MEP) in mmH2O
Respiratory flow performance | up to 3 weeks
  peak inspiratory (PIFR) and expiratory flows (PEFR) in liter per minute

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hogg JC. Lung structure and function in COPD. Int J Tuberc Lung Dis. 2008 May;12(5):467-79. PMID 18419881
- [Background] Hogg JC, Timens W. The pathology of chronic obstructive pulmonary disease. Annu Rev Pathol. 2009;4:435-59. doi: 10.1146/annurev.pathol.4.110807.092145. PMID 18954287
- [Background] Baraldo S, Turato G, Saetta M. Pathophysiology of the small airways in chronic obstructive pulmonary disease. Respiration. 2012;84(2):89-97. doi: 10.1159/000341382. Epub 2012 Aug 6. PMID 22868355
- [Background] Barnes PJ, Celli BR. Systemic manifestations and comorbidities of COPD. Eur Respir J. 2009 May;33(5):1165-85. doi: 10.1183/09031936.00128008. PMID 19407051
- [Background] Rossi A, Ganassini A, Polese G, Grassi V. Pulmonary hyperinflation and ventilator-dependent patients. Eur Respir J. 1997 Jul;10(7):1663-74. doi: 10.1183/09031936.97.10071663. PMID 9230263
- [Background] Gagnon P, Guenette JA, Langer D, Laviolette L, Mainguy V, Maltais F, Ribeiro F, Saey D. Pathogenesis of hyperinflation in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Feb 15;9:187-201. doi: 10.2147/COPD.S38934. eCollection 2014. PMID 24600216
- [Background] Krieger BP. Hyperinflation and intrinsic positive end-expiratory pressure: less room to breathe. Respiration. 2009;77(3):344-50. doi: 10.1159/000192790. Epub 2009 Jan 10. PMID 19141987
- [Background] Langer D, Ciavaglia CE, Neder JA, Webb KA, O'Donnell DE. Lung hyperinflation in chronic obstructive pulmonary disease: mechanisms, clinical implications and treatment. Expert Rev Respir Med. 2014 Dec;8(6):731-49. doi: 10.1586/17476348.2014.949676. Epub 2014 Aug 27. PMID 25159007
- [Background] O'Donnell DE, Webb KA, Neder JA. Lung hyperinflation in COPD: applying physiology to clinical practice. COPD Res Pract. 2015;1(1):4
- [Background] O'Donnell DE, Laveneziana P. Physiology and consequences of lung hyperinflation in COPD. Eur Respir Rev. 2006;15(100):61-67
- [Background] Somfay A, Porszasz J, Lee SM, Casaburi R. Dose-response effect of oxygen on hyperinflation and exercise endurance in nonhypoxaemic COPD patients. Eur Respir J. 2001 Jul;18(1):77-84. doi: 10.1183/09031936.01.00082201. PMID 11510809
- [Background] Spahija J, Marchie Md, Ghezzo H, Grassino A. Factors discriminating spontaneous pursed-lips breathing use in patients with COPD. COPD. 2010 Aug;7(4):254-61. doi: 10.3109/15412555.2010.496820. PMID 20673034
- [Background] Gigliotti F, Coli C, Bianchi R, Romagnoli I, Lanini B, Binazzi B, Scano G. Exercise training improves exertional dyspnea in patients with COPD: evidence of the role of mechanical factors. Chest. 2003 Jun;123(6):1794-802. doi: 10.1378/chest.123.6.1794. PMID 12796152
- [Background] Puente-Maestu L, Stringer WW. Hyperinflation and its management in COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(4):381-400. doi: 10.2147/copd.2006.1.4.381. PMID 18044095
- [Background] Ichiba T, Miyagawa T, Kera T, Tsuda T. Effect of manual chest wall compression in participants with chronic obstructive pulmonary disease. J Phys Ther Sci. 2018 Nov;30(11):1349-1354. doi: 10.1589/jpts.30.1349. Epub 2018 Nov 6. PMID 30464362
- [Background] Nozoe M, Mase K, Ogino T, Murakami S, Takashima S, Domen K. Effects of chest wall compression on expiratory flow rates in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2016 Mar 15;20(2):158-65. doi: 10.1590/bjpt-rbf.2014.0145. PMID 26982453
- [Background] Mase K, Yamamoto K, Murakami S, Kihara K, Matsushita K, Nozoe M, Takashima S. Changes in ventilation mechanics during expiratory rib cage compression in healthy males. J Phys Ther Sci. 2018 Jun;30(6):820-824. doi: 10.1589/jpts.30.820. Epub 2018 Jun 12. PMID 29950772
- [Background] Brunherotti MA, Martinez FE. Response of oxygen saturation in preterm infants receiving rib cage stabilization with an elastic band in two body positions: a randomized clinical trial. Braz J Phys Ther. 2013 Mar-Apr;17(2):105-11. doi: 10.1590/S1413-35552012005000082. English, Portuguese. PMID 23778773
- [Background] Celli B, Fabbri L, Criner G, Martinez FJ, Mannino D, Vogelmeier C, Montes de Oca M, Papi A, Sin DD, Han MK, Agusti A. Definition and Nomenclature of Chronic Obstructive Pulmonary Disease: Time for Its Revision. Am J Respir Crit Care Med. 2022 Dec 1;206(11):1317-1325. doi: 10.1164/rccm.202204-0671PP. No abstract available. PMID 35914087
- [Background] Pellegrino R, Brusasco V. On the causes of lung hyperinflation during bronchoconstriction. Eur Respir J. 1997 Feb;10(2):468-75. doi: 10.1183/09031936.97.10020468. PMID 9042651
- [Background] De Troyer A. Effect of hyperinflation on the diaphragm. Eur Respir J. 1997 Mar;10(3):708-13. PMID 9073010
- [Background] Decramer M. Hyperinflation and respiratory muscle interaction. Eur Respir J. 1997 Apr;10(4):934-41. PMID 9150337
- [Background] Munari AB, Venancio RS, Gulart AA, Da Silveira JA, Klein SR, Martins AC, Mayer AF. Slow chest compression acutely reduces dynamic hyperinflation in people with chronic obstructive pulmonary disease: a randomized cross-over trial. Physiother Theory Pract. 2022 Dec;38(12):1937-1945. doi: 10.1080/09593985.2021.1907824. Epub 2021 Apr 8. PMID 33829946